CLINICAL TRIAL: NCT02629406
Title: Studies on the Adaptive Responses (Cardiovascular, Respiratory and Angiogenetic) to Hypoxia in Patients With Type 1 Diabetes Compared to Controls
Brief Title: Studies on the Adaptive Responses to Hypoxia
Acronym: HYKRAND
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Neda Rajamand Ekberg, M.D, PhD, Karolinska University Hospital
Other Study IDs: 2015/1182-31/4.
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Hypoxia; Diabetes Mellitus, Type 1
Keywords: HIF; hypoxia; chemoreflex; baroreflex; MIR210
MeSH Terms: conditions — Hypoxia; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Diabetes typ 1: Patients with typ 1diabetes with a duration of the disease between 10-20 years (HbA1C >65 mmol/l) and age 20-50 will be exposed to intermittent hypoxia.
  Interventions: Other: Hypoxia
- Healthy controls: Healthy controls, age 20-50 will be exposed to intermittent hypoxia.
  Interventions: Other: Hypoxia

INTERVENTIONS:
Other: Hypoxia — Intermittent hypoxia which consist of five hypoxic periods (13% O2 inspired fraction of oxygen) each lasting 6 min, with five normoxic intervals of same duration

SUMMARY:
The general aim of this study is to define the response to hypoxic challenge in patients with diabetes. The investigation will provide response for different questions that are central for explaining the development of complications in diabetes

* have patients with diabetes an impaired reaction to adapt to hypoxia
* what consequence has hypoxia challenge on respiratory and on cardiovascular regulation in patients with diabetes
* what consequence has diabetes on the angiogenetic response to hypoxia

DETAILED DESCRIPTION:
Complications of diabetes represent the main concern for modern diabetes therapy, and it has become a priority to further characterise the pathophysiological mechanisms of these complications to ensure the development of novel rational therapeutic strategies.

Although the prolonged exposure of tissues to hyperglycaemia is the primary causative factor for chronic diabetes complications, it has recently become increasingly evident that hypoxia also plays an important role in all diabetes complications . A low tissue concentration of oxygen in diabetes is the consequence of several mechanisms (e.g., deficient blood supply because of micro- and macro-vascular disease , poor local oxygen diffusion because of local oedema, or as the result of increased oxygen consumption).

Adaptive responses of cells to hypoxia are mediated by Hypoxia-Inducible Factor 1 (HIF), which is a heterodimeric transcription factor that is composed of and subunits, which are both constitutively expressed in mammalian cells. The regulation of HIF activity is critically dependent on subunit degradation in normoxia. Under hypoxic conditions, HIF-1 is stabilised, binds to HRE (hypoxic responsive elements) and up-regulates a gene series that is involved in angiogenesis, glycolytic energy metabolism, cell proliferation, and survival, which enables cells to adapt to reduced oxygen availability. It is estimated that that more than 800 genes are direct HIF targets . HIF-1 is central for expression of multiple angiogenic growth factors (reviewed by[6]), endothelial progenitor cells (EPC) recruitment . Recently, it has been proposed that microRNAs (ex. mir210) also mediate some HIF-1 functions .

Several pieces of evidence point to a defective response of diabetic tissues to hypoxia. An impaired hypoxia response is present in all tissues investigated in diabetic animal and diabetic patients. Hyperglycaemia directly represses HIF stability and function at multiple levels, a mechanism that is not completely understood.

An impaired reaction to hypoxia in diabetes might have important consequences in acute hypoxic challenges as acute heart infarction, stroke, limb ischemia but also in subtle regulation of cardiovascular and respiratory system as a consequence of autonomic neuropathy with potential severe prognostic effect on late cardiovascular events . Interventional studies have addressed the cardiovascular responses to intermittent hypoxia (IH) compared with normoxia exposure in patients with diabetes . However in order to establish the appropriateness of the cardiovascular reaction to hypoxia in diabetes it is a need to investigate the cardiorespiratory responses towards IH in patients with diabetes compared with matched non diabetic control subjects. Moreover it is essentially to establish the angiogenetic response in the same experimental design. The hypothesis for this study is that both the cardiorespiratory reaction mediated through autonomic nervous system and angiogenetic response are impaired in patients with diabetes as a consequence of an impaired HIF reaction as seen in other tissues .

The investigators plan to study the effect of intermittent hypoxia (IH) that will consists of five hypoxic periods (13% O2 inspired fraction of oxygen) each lasting 6 min, with five normoxic intervals of same duration in 15 patients with type 1 diabetes without clinical signs of neuropathy and in 15 non diabetic controls matched for sex, BMI, age. The study will be performed during one day.

Methods:

Baseline data will be obtained in the morning of each testing day at least 2 h after breakfast. Subjects are advised to abstain from caffeinated beverages for 12 h and from alcohol for 36 h prior to testing.

Blood pressure and heart rate and arterial oxygen saturation will be continuously measured. In case of a decrease in oxygen saturation 80% or the occurrence of symptoms, hypoxia would have been discontinued until oxygen levels reached at least 80%. A technician will regulate and control the breathing periods under supervision of a medical doctor in a way that the intervention could not be observed by any patient. Thereafter, three measurement sessions will be performed: immediately after (t2), after 3 h (t3), and after 6 h (t4). After t2, each patient will obtaine an individual meal according to diet requirement.

Cardiovascular and respiratory testing.

Hypoxic ventilatory response (HVR) and hypercapnic ventilatory response (HCVR) will be evaluated to determine respiratory system activity. All patients will be tested in the supine position in a silent room at comfortable temperature. Before participants will be connected to a rebreathing circuit through a mouthpiece with an antibacterial filter, spontaneous breathing of room air at rest will be performed for4 min in order to obtain baseline data.

During each condition, the investigators will perform continuous measurement of oxygen saturation (SaO2) by a pulse oximeter and end-tidal CO2 (CO2-et) using a capnograph connected to a mouthpiece. Recordings of electrocardiogram will be performed by chest leads, and continuous noninvasive blood pressure will be recorded using the cuff method. A heated Fleish pneumotachograph will be connected to a differential pressure transducer and inserted in series to the expiratory component of the rebreathing system to measure airway flow. For measurement of the response to hypoxia, the participants will be connected to a rebreathing circuit inducing progressive decrease in SaO2 while maintaining CO2-et values at constant levels, until SaO2 will reach 80%, and measuring breath-to-breath changes in minute ventilation. The response to hypercapnia will be evaluated by ventilatory changes induced by progressive increase in CO2-et levels (up to 13 mmHg above resting levels), while SaO2 will be maintained 98% by oxygen at very low flow.

Cardiovascular autonomic function will be determined performing four tests according to recent guidelines: deep-breathing, 30:15 ratio, Valsalva maneuver and systolic blood pressure response to standing. Cardiovascular autonomic neuropathy will be defined as the "presence of two or more abnormal tests".

Measurement of chemoreflex sensitivity: The slope of the linear regression line of minute ventilation versus SaO2 or CO2-et indicates in each case the chemoreflex sensitivity to hypoxia or hypercapnia. In the hypercapnic test, the point at which the ventilation start to increase indicates as ventilator recruitment threshold to CO2 (VRT- CO2). VRT- CO2 will be identified by interpolating the ventilation/CO2-et plot by a fourth-order polynomial function.

Assessment of baroreflex sensitivity: The baroreflex sensitivity (BRS) will be measured during spontaneous breathing at each measurement session. Since previous studies did not document a better performance of one method over the others, the investigators will calculate the average of seven different methods: positive and negative sequences, the a-coefficient in the low- and high-frequency bands and its average, the transfer function technique, and the ratio of SDs of R-R interval and systolic blood pressure variabilities. Besides BRS, SD of the R-R interval (SDNN) will be applied to determine a global index of heart rate variability. This selection is done based on the fact that normal distribution is more pronounced in this variable compared with other indices of variability (e.g., variance). The Hypoxic ventilatory response (HVR) and hypercapnic ventilatory response (HCVR), baroreflex sensitivity (BRS) will be evaluated before (t1), immediately after (t2), 3 h (t3), and 6 h (t4) after IH.

The angiogenetic potential will be evaluated at the same endpoints by measuring in serum relevant cytokines that are gene targets for HIF-1 (i.e. VEGFA, SDF-1a, erythropoietin etc). The direct response of HIF signaling will be evaluated by the serum levels of mir210 which exclusively regulated by HIF.

The absolute endothelial precoursor cell account (EPC) response will be evaluated at the same time points by FACS analysis of the number of CD34+/CD133+/KDR +

ELIGIBILITY:
Inclusion Criteria:

1. Patients with typ1 diabetes with a duration of the disease between 10-20 years (HbA1c ≥ 65 mmol /l)
2. Healthy controls matched for age, BMI and gender on group bases.

Exclusion Criteria:

1. Smoking
2. Infections during the last month
3. Major cardiovascular complications such as coronary heart disease, unstable or stable angina, myocardial infarction, ventricular arrhythmias, and atrial fibrillation in the last 3 months
4. Decompensated congestive heart failure or functional class 3-4.
5. Therapy with b-blockers
6. Severe hypertension (180 mmHg systolic or 110 mmHg diastolic blood pressure
7. Proliferative retinopathy.
8. Obvious sign for diabetic neuropathy (decreased/absent sensitivity to 10 g monofilament, vibration, plantar reflex)
9. Definite autonomic dysfunction
10. HbA1c ≥ 108 mmol/l
11. Any concomitant disease or condition that may interfere with the possibility for the patient to comply with or complete the study protocol
12. Malignancy
13. History of alcohol or drug abuse
14. Participant in another ongoing pharmacological study
15. Unwillingness to participate following oral and written information
16. Subjects with any other severe acute or chronic medical or psychiatric condition that make the subject inappropriate for the study in the judgment of the investigator

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with diabetes are included from Department of endocrinology. Healthy controls are included via announcement och social media.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-11; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Endothelial precursor cell account (EPC) | 24 hours
  The absolute amount of endothelial precursor cells in 10 ml of blood

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Catrina, ass. prof., Principal Investigator — Karolinska Institutet, Stockholm, 17176, Sweden
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden